CLINICAL TRIAL: NCT00166465
Title: A Phase I Dose-Finding Study and a Randomized Phase II Study of ALIMTA Plus Oxaliplatin Versus Oxaliplatin Plus 5-Fluorouracil and Leucovorin (FOLFOX 4 Regimen) in the First-Line Treatment of Patients With Locally Advanced Unresectable or Stage IV Colorectal Cancer
Brief Title: Stage IV Colorectal CA ALIMTA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Steven R. Alberts, M.D., Mayo Clinic Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0248; MC0248 (Other: Mayo Clinic Cancer Center); 1126-03 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Locally Advanced Unresectable or Stage IV Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ALIMTA plus Oxaliplatin versus Oxaliplatin plus 5-Fluorouracil and Leucovorin (FOLFOX 4 Regimen)

SUMMARY:
Phase I: The primary objective of the Phase 1 portion of this study is to determine the Maximum tolerated dose and the recommended Phase 2 dose of ALIMTA plus oxaliplatin when given with folate and vitamin B-12 supplementation in the treatment of patients with unresectable, locally advanced or metastatic colorectal cancer. The Phase I component of the study will be activated for enrollment of Mayo Clinic patients only.

Phase II: The primary objective of the Phase 2 portion of this study is to determine the tumor response rates to ALIMTA plus oxaliplatin and oxaliplatin plus 5-fluorouracil and leucovorin in patients with locally advanced unresectable or Stage IV colorectal cancer that have not received prior chemotherapy for advanced disease. Patients will be randomly assigned to receive either ALIMTA plus oxaliplatin (Arm A) or Oxaliplatin plus 5-Fluorouracil and Leucovorin (Arm B). The Phase II component of the study will be activated for enrollment of patients via the Mayo Clinic Cancer Research Consortium mechanism. A comparison will be made of the side effects between regimens.

DETAILED DESCRIPTION:
ALIMTA, oxaliplatin, and 5-fluorouracil (alone or with leucovorin) have shown activity as single agents in the treatment of colorectal cancer. Their different mechanisms of action make the combination of ALIMTA with oxaliplatin attractive as potential first-line therapies in terms of improving response rates and overall survival in patients with metastatic colorectal cancer. Current reports of the combination of oxaliplatin and 5-FU as first-line therapies suggest that there may be advantages in combining oxaliplatin with other antifolates in the treatment of colorectal cancer. ALIMTA is an attractive candidate to replace other drugs such as 5-FU in the combinations with oxaliplatin in the treatment of locally advanced and metastatic colorectal cancer. ALIMTA has potential advantages over 5-FU when combined with oxaliplatin because it requires a single short injection and inhibits multiple targets in the folate pathway. Therefore, we propose to conduct a trial reporting the clinical effectiveness and side effects of ALIMTA plus oxaliplatin and one of the current standards of care, the FOLFOX 4 regimen (Oxaliplatin plus 5-Fluorouracil and Leucovorin).

ELIGIBILITY:
Inclusion criteria

3.11 Phase I and II Required Characteristics

3.111 Pathologic or cytologic diagnosis of adenocarcinoma of the colon or rectum. Patients must have locally advanced unresectable or Stage IV colorectal cancer that is not amenable to curative therapy. See Protocol Appendix VI, American Joint Committee on Cancer Staging Criteria for Colorectal Cancer.

3.112 Measurable disease as defined by RECIST criteria (see Section 11.0). Patients who do not have measurable disease, but who do have evaluable disease, may be enrolled in the Ph I portion of the study only.

3.113 Prior radiation therapy allowed to <25% of the bone marrow (see Protocol Appendix VII, Distribution of Active Bone Marrow in the Adult), and patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Patients are allowed to have received standard postoperative adjuvant radiation therapy for rectal cancer. Prior radiotherapy must be completed < 30 days before study entry. Lesions that have been radiated in the advanced setting cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.

3.114 ECOG performance status (PS) of 0, 1or 2 (see Protocol Appendix IV).

3.115 Estimated life expectancy of greater than or equal to 12 weeks.

3.116 Ability and willingness to comply with adequate follow-up.

3.117 Adequate organ function including the following less than or equal to 7 days prior to study entry:

* Adequate bone marrow reserve:
* ANC greater than or equal to 1500
* PLT greater than or equal to 100,000
* Hgb greater than or equal to 9 g/dL.
* Hepatic:
* Total bilirubin less than or equal to 1.5 x ULN
* Alk Phos (AP), AST less than or equal to 3.0 x ULN (AP and AST less than or equal to 5 ULN is acceptable if liver has tumor involvement).
* Renal: calculated creatinine clearance (CrCl) >= 45 mL/min based on the standard Cockcroft and Gault formula (see table below) or on measured glomerular filtration rate (GFR) using the appropriate radiolabeled method (51-CrEDTA or Tc99m-DTPA). Enrollment and dosing decisions based on creatinine clearance may be made using local lab values (calculated using the standard Cockcroft and Gault formula [see below]) The serum creatinine must be assayed at the same local lab each time for that patient.

  * Cockcroft and Gault Equation Creatinine clearance for males = (140 - age)(weight in kg) (72)(serum creatinine in mg/dL) Creatinine clearance for females = 140 - age)(weight in kg)(0.85) (72)(serum creatinine in mg/dL) Moderate renal impairment is calculated creatinine clearance 30-50 mL/min (32). Mild renal impairment is calculated creatinine clearance 51-80 mL/min (32).

3.118 Ability to sign informed consent.

3.119 Age greater than or equal to 18 years.

Exclusion criteria

3.12 Phase I and II Contraindications

3.121 Evidence of peripheral neuropathy >CTCAE v3.0 Grade 1 (for example, diabetic neuropathy).

3.122 Prior chemotherapy for advanced disease. Only one prior adjuvant therapy including CPT-11, or 5-fluorouracil-leucovorin, Capecitabine but not oxaliplatin is allowed if it has been >= 6 months since the last treatment. Patients enrolling in the Phase I portion of the trial may have received one advanced disease regimen that does not include either ALIMTA or oxaliplatin.

3.123 Treatment less than or equal to 30 days with any chemotherapy as well as non-cytotoxic cancer therapy such as immunotherapy.

3.124 Serious concomitant systemic disorders (including active infections or uncontrolled/brittle diabetes) that would compromise the safety of the patient or compromise the patients ability to complete the study.

3.125 Second primary malignancy (except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated >= 5 years previously with no evidence of recurrence; prior low grade [Gleason score £ 6] localized prostate cancer is allowed).

3.126 Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents 2 days before, the day of, and 2 days after each dose of ALIMTA (5 days prior for long-acting agents such as piroxicam). (See Appendix VIII for list of NSAIDs.)

3.127 Clinically symptomatic central nervous system metastases. Metastases that have been previously treated and are stable are allowed as judged by the investigator.

3.128 Any of the following as this regimen may be harmful to a developing fetus or nursing child:

* Pregnant women
* Nursing women
* Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device (IUD), surgical sterilization, subcutaneous implants, or abstinence, etc.)

3.129a Presence of clinically relevant third-space fluid collections. Fluid collections may be drained to allow the patient to enroll in the study.

3.129b Weight loss ³10% - 6 weeks prior to study entry.

3.129c Inability or unwillingness to take folic acid or vitamin B12.

3.129d Previous completion or withdrawal from this study or any other study investigating ALIMTA.

3.129e Prior treatment with oxaliplatin.

3.129f Concurrent therapy or treatment - 30 days with another experimental agent for cancer or other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated using the exact binomial distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States